CLINICAL TRIAL: NCT07308054
Title: The Effects of Fresnel Prism Glasses on Visual Perception, Balance, Gait and Functional Independence in Post-Stroke Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore University of Biological and Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UBAS/ERB/FpRS/25/035
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Stroke
Keywords: Visual Perception; Functional Independence; Fresnel Prism Glasses; Gait; Balance
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: After recruitment of participants into the study, they will be allocated to their respective group utilizing the online randomization tool.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm/group (Experimental): Participants allocated to the experimental group will receive Fresnel prism glasses (15 prism diopters) in addition to conventional physiotherapy. The Fresnel prism lenses will be affixed to the participant's spectacles to induce visuospatial realignment during therapeutic activities. Participants will wear the prism glasses during supervised rehabilitation sessions focused on balance training, gait training, and functional mobility tasks. Conventional physiotherapy will include postural control exercises, weight-shifting activities, gait re-education, and task-oriented functional training. The intervention will be administered for 4 weeks, with sessions conducted 5 days per week, under the supervision of a qualified physiotherapist.
  Interventions: Device: Fresnel Prism Glasse; Behavioral: Convetional physical therapy
- Arm/Group (Active Comparator): Participants allocated to the control group will receive conventional physiotherapy alone, without the use of Fresnel prism glasses. The rehabilitation program will follow standard neurorehabilitation protocols and will include balance exercises, gait training, strengthening, postural alignment exercises, and functional mobility tasks. Therapy will be provided with the same frequency and duration as the experimental group (5 sessions per week for 4 weeks) to ensure comparability between groups.
  Interventions: Behavioral: Convetional physical therapy

INTERVENTIONS:
Device: Fresnel Prism Glasse — Fresnel prism glasses consist of lightweight, flexible, press-on plastic prism lenses with a power of 15 prism diopters, affixed to the inner surface of standard spectacle lenses. The prisms are designed to shift the visual field horizontally to promote visuospatial realignment and improve sensory integration during functional activities.
  Participants assigned to the experimental group will wear Fresnel prism glasses during supervised physiotherapy sessions. The intervention will be administered alongside conventional physiotherapy, including balance training, gait training, postural control exercises, and functional mobility tasks. The prism glasses will be worn throughout the therapy session to facilitate visual feedback and encourage symmetrical weight-bearing and improved postural alignment.
  The intervention will be delivered for a duration of 4 weeks, with sessions conducted 5 days per week. Each session will last approximately 30-45 minutes and will be supervised by a qualified
Behavioral: Convetional physical therapy — Conventional physiotherapy will be provided to all participants in both groups according to standard neurorehabilitation protocols. The program will include balance exercises, gait training, strengthening exercises, postural alignment activities, weight-shifting exercises, and task-oriented functional training. Participants in the control group will receive conventional physiotherapy alone, without Fresnel prism glasses, for the same duration and frequency as the experimental group.

SUMMARY:
This randomized controlled trial aims to evaluate the effects of Fresnel prism glasses on visual perception, balance, gait, and functional independence in post-stroke patients. Stroke survivors, particularly those with right hemisphere involvement, often experience visuospatial deficits such as unilateral spatial neglect, leading to impaired balance, abnormal gait, and reduced functional independence. Fresnel prism glasses offer a low-cost, non-invasive intervention that may improve visuospatial alignment and postural control by modifying visual input. Adult post-stroke patients will be randomly allocated into an intervention group receiving Fresnel prism glasses alongside conventional physical therapy, and a control group receiving conventional therapy alone. Outcome measures will include the Motor-Free Visual Perception Test, Berg Balance Scale, Functional Independence Measure, and JAKC Observational Gait Analysis. Assessments will be conducted at baseline, post-intervention, and follow-up. The study is expected to provide evidence on whether Fresnel prism glasses can serve as an effective adjunct to conventional rehabilitation for improving mobility, balance, and functional outcomes in stroke survivors.

DETAILED DESCRIPTION:
Stroke is one of the leading causes of long-term disability worldwide and is frequently associated with impairments in balance, gait, motor function, and visuospatial perception. Among these deficits, unilateral spatial neglect (USN) is particularly common following right hemisphere stroke and significantly limits functional recovery. Individuals with USN often demonstrate impaired awareness of the contralesional space, distorted midline perception, postural asymmetry, and abnormal gait patterns, which collectively increase the risk of falls and dependence in activities of daily living. Despite advances in conventional stroke rehabilitation, including physical and occupational therapy, many patients continue to experience persistent functional limitations, highlighting the need for innovative and adjunctive rehabilitation strategies.

Recent developments in neurorehabilitation emphasize sensory-based interventions that promote neuroplasticity by modifying sensory input. Fresnel prism glasses represent a low-cost, non-invasive visual intervention designed to shift the visual field and facilitate visuospatial realignment. By altering visual input, Fresnel prisms may enhance sensory integration and improve postural control, balance, and gait performance in stroke survivors. Preliminary studies have demonstrated improvements in balance measures, gait symmetry, and visual perception following prism use; however, findings remain inconsistent, and evidence regarding functional outcomes and long-term effects is limited.

This randomized controlled trial aims to evaluate the effectiveness of Fresnel prism glasses as an adjunct to conventional physiotherapy in post-stroke patients. Eligible participants with a confirmed diagnosis of stroke will be randomly allocated into two groups: an experimental group receiving Fresnel prism glasses in addition to standard rehabilitation, and a control group receiving conventional physiotherapy alone. The intervention will be delivered over a defined treatment period, with assessments conducted at baseline and post-intervention.

Primary outcome measures will assess balance and postural control using standardized tools such as the Berg Balance Scale and Functional Reach Test. Secondary outcomes will include gait analysis, visual perception, and functional independence measured through validated clinical scales. The study also seeks to examine whether visual realignment through Fresnel prisms can facilitate weight transfer toward the affected side and reduce asymmetry during standing and walking.

The findings of this study are expected to contribute to the growing body of evidence on sensory-based rehabilitation interventions for stroke. By addressing current gaps related to functional outcomes and feasibility, this research may help establish Fresnel prism glasses as an effective, accessible adjunct therapy in stroke rehabilitation, particularly in resource-limited settings. Ultimately, the study aims to support improved mobility, independence, and quality of life among stroke survivors.

ELIGIBILITY:
Inclusion Criteria Right hemisphere with left side neglect (14). Adults (40-65 years old) who have experienced an ischemic stroke for the first time (1-3 months post-stroke) are eligible (15) A score of 2-4 in the Functional Ambulation Category (FAC) (16) and MMSE ≥24 (to guarantee training-related cognitive ability)(17). Patient who can walk more than 10m Independently Exclusion Criteria Severe comorbidities, such as neurological or orthopedic disorders and impair gait(18) Hearing and vision problems that are not assisted. Patients with profound sensory impairment or significant cognitive dysfunction(19) Individuals who have recently suffered from cardiac failure, myocardial infarction, or other severe illnesses(20)

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-13 (Estimated); Primary Completion 2026-05-26 (Estimated); Study Completion 2026-05-26 (Estimated)

PRIMARY OUTCOMES:
Motor-Free Visual Perception Test | Baseline, before intervention, 8 weeks post intervention
  The Motor-Free Visual Perception Test (MVPT) is a standardized assessment tool consisting of 36 items that evaluate multiple domains of visual perception, including figure-ground discrimination, visual discrimination, visual memory, visual closure, and spatial relationships. It is designed to assess visual field deficits and overall visual perceptual function in patients who have experienced brain injuries or strokes. In this study, we measured participants' response behaviors to identify the extent of unilateral neglect by recording their responses to both the left and right sides of the body, regardless of accuracy. Correct responses are scored as raw points, while the total time taken to complete the assessment is recorded as the visual perceptual processing time. The maximum score achievable is 36 points. The MVPT demonstrates high reliability, with a test-retest intraclass correlation coefficient (ICC) of 0.92 (95% CI: 0.84-0.96). In this trial, the MVPT will be utilized.
Berg Balance Scale | baseline, before interventio, 8 weeks post intervention
  The Functional Independence Measure (FIM) is a key tool used to assess the level of disability in patients undergoing rehabilitation. It evaluates 18 different activities of daily living on a scale from 1 to 7, where 1 means the person is fully dependent and 7 means they can do everything independently without any assistance. The highest possible score is 126, which signifies complete functional independence, while the lowest score of 18 indicates total dependence. The activities are divided into two main categories: 13 motor skills (like personal care, sphincter control, mobility, and locomotion) and five cognitive skills (which include communication and social cognition)
Functional Independence Measure | baseline, before intervention, 8 weeks post intervention
  Independence Measure (FIM) is a key tool used to assess the level of disability in patients undergoing rehabilitation. It evaluates 18 different activities of daily living on a scale from 1 to 7, where 1 means the person is fully dependent and 7 means they can do everything independently without any assistance(23). The highest possible score is 126, which signifies complete functional independence, while the lowest score of 18 indicates total dependence. The activities are divided into two main categories: 13 motor skills (like personal care, sphincter control, mobility, and locomotion) and five cognitive skills (which include communication and social cognition)
JAKC's Observational Gait Analysis | Baseline, before intervention, 8 week post intervention
  The JAKC Observational Gait Analysis (Joint Angle Kinematic Coordination) is a wellstructured clinical tool designed to evaluate gait patterns, especially in individuals dealing with neurological or musculoskeletal issues like stroke. It zeroes in on the coordination and quality of movement in key joints-namely the hip, knee, ankle, and trunk-throughout various stages of the gait cycle. By closely observing joint angles, timing, and how limbs work together, therapists can spot unusual movement patterns and compensatory behaviors. The JAKC scale aids in clinical decision-making by pinpointing specific gait deviations, which helps in crafting targeted interventions and tracking progress over time. It's a practical, non-invasive approach that's widely embraced in rehabilitation environments

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ha SY, Sung YH. Effects of Fresnel prism glasses on balance and gait in stroke patients with hemiplegia: A randomized controlled trial pilot study. Technol Health Care. 2020;28(6):625-633. doi: 10.3233/THC-191973. PMID 32280072